CLINICAL TRIAL: NCT01742897
Title: Evaluation of Efficacy and Safety of TTS-Fentanyl in Moderate to Severe Pain From Knee Osteoarthritis
Brief Title: Efficacy and Safety Study of Transdermal Therapeutic System (TTS) Fentanyl in Participants With Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014524; FENPAI4052
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Transdermal therapeutic system (TTS) fentanyl; Durogesic
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TTS-fentanyl (Experimental): Transdermal therapeutic system (TTS) fentanyl patches releasing at the rate of 12.5 microgram per hour for 3 days. The patches will be replaced every 3 days until 30 days.
  Interventions: Drug: TTS-fentanyl

INTERVENTIONS:
Drug: TTS-fentanyl
  Other Names: Durogesic

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Transdermal therapeutic system (TTS) fentanyl patches (transdermal patch containing a drug that is put on the skin so the drug will enter the body through the skin) in knee osteoarthritis (disorder, which is seen mostly in older persons, in which the joints become painful and stiff) participants with moderate to severe pain.

DETAILED DESCRIPTION:
This is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), single-arm, prospective study (study following participants forward in time) of TTS-fentanyl matrix form in knee osteoarthritis participants. The study consists of 3 phases: a screening phase, an open label treatment phase consisting of 2 periods, and an evaluation phase. The first patch will be applied on the first day of treatment phase by the investigator, and sufficient patches until Day 30 will be provided to the participant with the instructions to apply the patch. The TTS-fentanyl dose will normally be increased, if needed by 12.5 microgram per hour taking into account the daily dose of supplemental paracetamol required by the participant. Efficacy with regard to pain control will be recorded principally by the participant via questionnaires in a daily diary. This record will be used to support more detailed assessments at study visits on Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire. Participants' safety will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (lasting a long time) primary osteoarthritis knee pain, one or two side with stage II Kellgen-Lawrence, for more than 3 months with Visual Analogue Scale (VAS) more than 4
* Good knee deformity, no limit range of motion
* Participant who has signed the informed consent form

Exclusion Criteria:

* Skin disease that prevents the use of the transdermal system or which could affect the absorption of fentanyl or local tolerability
* History or suspicion of alcohol or drug abuse within the past 5 years
* History of cardiac, nervous system or respiratory disease which in the investigator's judgment prevents participation in the study because of the potential for respiratory depression
* Confusion, reduced level of consciousness, or concomitant psychiatric disorder which, in the opinion of the investigator, could prevent participation in the trial
* Participants who do not understand or speak Thai

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd., Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (1):
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- TTS-Fentanyl: Transdermal therapeutic system (TTS) fentanyl patches releasing at the rate of 12.5 microgram per hour for 3 days. The patches were replaced every 3 days until 30 days.
Period: Overall Study
Arm/Group | TTS-Fentanyl
Started | 35
Treated | 33
Completed | 30
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | TTS-Fentanyl
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: Years] | 66.34 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 1
Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) Scores [Mean (Standard Deviation); unit: Millimeter (mm)] — The WOMAC is a self administered, participant health related questionnaire consisting of three subscales (pain, stiffness and physical function). Pain subscale score ranges from 0-100 mm (0 mm=no pain to 100 mm=extreme pain); stiffness subscale score ranges from 0-100 mm (0 mm=no stiffness to 100 mm=extreme stiffness) and physical function subscale ranges from 0-100 mm (0 mm=no difficulty to 100 mm=extreme difficulty). The overall WOMAC score is the sum of the 3 subscale scores which ranges from 0-300 mm (0 mm=none to 300 mm=extreme/worst).
  Millimeter (mm)
    Pain | 43.9 (1.51)
    Stiffness | 41.6 (1.92)
    Physical function | 47.6 (1.12)
    Overall | 133.1 (4.04)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) Score at Day 30
Description: The WOMAC is a self administered, participant health related questionnaire consisting of three subscales (pain, stiffness and physical function). Pain subscale score ranges from 0-100 mm (0 mm=no pain to 100 mm=extreme pain); stiffness subscale score ranges from 0-100 mm (0 mm=no stiffness to 100 mm=extreme stiffness) and physical function subscale ranges from 0-100 mm (0 mm=no difficulty to 100 mm=extreme difficulty). The overall WOMAC score is the sum of the 3 subscale scores which ranges from 0-300 mm (0 mm=none to 300 mm=extreme/worst).
Time Frame: Baseline, Day 30
Population: Intent-to-treat (ITT) analysis population included all participants regardless of their compliance with the protocol.
Measure: Median (95% Confidence Interval); unit: Millimeter (mm)
Arm/Group | TTS-Fentanyl
Number analyzed (Participants) | 35
Millimeter (mm)
  Pain | -22.2 [-28.42 to -15.97]
  Stiffness | -21.5 [-28.66 to -14.26]
  Physical function | -29.5 [-34.06 to -24.93]
  Overall | -73.2 [-88.63 to -57.67]

ADVERSE EVENTS:
Arm/Group | TTS-Fentanyl
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 10/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TTS-Fentanyl (N=33)
Nausea (General disorders) | 7
Vomiting (General disorders) | 7
Dizziness (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Company shall have right to publish data or information generated in trial without approval of Principal Investigator (PI). PI shall have right to publish results and information provided by Company if necessary. Prior to submission, PI will provide company 60 days for review. No paper with confidential Information will be submitted without company consent. If requested, PI will withhold it for 60 days to allow patent application filing. PI warrants compliance of all personnel involved in Study.